CLINICAL TRIAL: NCT02260466
Title: AMYLO-CARTESIAN Study :Prevalence and Post-surgical Outcomes of CARdiac Wild-type TransthyrEtin amyloidoSIs in Elderly Patients With Aortic steNosis Referred for Valvular Replacement.
Brief Title: Prevalence and Post-surgical Outcomes of CARdiac Wild-type TransthyrEtin amyloidoSIs in Elderly Patients With Aortic steNosis Referred for Valvular Replacement.
Acronym: AMYLOCARTESIAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Pfizer (Industry); Henri Mondor University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2013-02
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Heart Disease; Aging; Amyloidosis; Aortic Valve Stenosis
Keywords: Amyloidosis; echocardiography; magnetic resonance imaging; radionuclide imaging
MeSH Terms: conditions — Heart Diseases; Amyloidosis; Aortic Valve Stenosis

ARMS (1):
- elderly patients with Aortic steNosis valvular replacement (Other)
  Interventions: Other: a basal LV septum biopsy

INTERVENTIONS:
Other: a basal LV septum biopsy — During surgery, a basal LV septum biopsy will be collected for determination and quantification of interstitial deposits using specific staining which will be performed in a blind fashion

SUMMARY:
Background: The prevalence of both senile cardiac amyloidosis (CA) and aortic stenosis (AS) markedly increases with age. Aortic stenosis increases left ventricular pressure overload. Cardiac deposits have been observed in AS and the amount of these deposits has been correlated to post-surgical outcome. As they are strong echocardiographic and cardiac MRI imaging similarities between CA and AS, the investigators hypothesized that the deposit observed in AS is transthyretin amyloid deposit. The investigators objective is to demonstrate that amyloid deposit is associated with poor outcomes following aortic stenosis surgical valve replacement.

Materiel and methods: 180 patients with indication for surgical aortic valve replacement will be recruited prospectively and consecutively in 5 French centers. A replicative study will be performed in one Austrian center. Echocardiography, cardiac MRI and bone scintigraphy will be performed prior to surgery. During surgery, a basal LV septum biopsy will be collected for determination and quantification of interstitial deposits using specific staining which will be performed in a blind fashion. Clinical outcomes will be recorded during the hospitalization period following the surgery and at 1 year. Alive and re-hospitalization status will be determined. Patients will be classified according to the presence or not of amyloid deposits.

Expected results and impact: This study will emphasize how pressure overload stress accelerates and magnifies amyloid deposition usually known to be related to cardiac aging process. It will develop reliable imaging tools and markers to detect cardiac amyloid deposition. Correlation between anatomopathologic analyses and the three different imaging technics will identify accurate imaging markers of CA. A risk stratification model based on amyloid deposits level for the clinical management of these patients will be created combining imaging and biological markers.

DETAILED DESCRIPTION:
Cardiovascular diseases remain the major cause of mortality and morbidity in industrialised countries. Their prevalence increases steeply as consequence of the aging of the population in these countries. Curiously, cardiovascular and neurodegenerative diseases share common aging pathological pathways involving abnormal accumulation of insoluble amyloid proteins in the extracellular matrix disrupting normal organ function. Whereas neurological amyloid diseases has been considerably investigated, little attention has been paid to the aggregation of amyloid proteins in cardiovascular diseases. Post-mortem studies have identified cardiac wild-type transthyretin amyloidosis deposition in 25% of individuals over the age of 80 years leading to the concept of "senile cardiac amyloidosis" (CA) (Cornwell, Am j Med 1984; Pitkanen, Am J Pathol 1984). The cause of this deposition is not yet known but might be related primarily to aging process and enhanced by cardiac mechanical stress (overload), hypoxia, oxidative stress and inflammation. Since patients with transthyretin CA develop severe heart failure with poor prognosis, it is crucial to identify them especially among population at risk such those with aortic stenosis (AS). Indeed this common valvular heart disease affects mainly senescent subjects and combines so the adverse effects on myocardial function of both pressure overload and myocardial aging.

Interestingly, some elderly patients with severe AS exhibit similar echocardiographic and cardiac MRI patterns as those reported in CA including increased cardiac wall thickness and progressive left ventricular dysfunction starting with alteration of basal LV-2D strain. They also exhibit increased late gadolinium enhancement (LGE) at cardiac MRI. This has been interpreted as related to interstitial myocardial "fibrosis" and has been correlated with poor prognosis after aortic valve replacement i.e.; high mortality, persistence of heart failure symptoms and LV dysfunction (Weidemann Circ 2009; Dweck, JACC 2011; Hermann JACC 2011). However none of these patients have benefited from a detailed histology analysis with aiming at identifying amyloid deposits. The investigators have recently found similar clinical observations in the investigators AS cohort. Using specific staining, the investigators were able to unmask the association of severe AS and CA in these patients. These preliminary findings raise the question of a potential pathophysiological link between CA and AS and might explain why some patients with AS may not benefit from cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Significant aortic stenosis. The aortic stenosis severity (aortic area : <1cm² or <0.6cm²/m² measured by echocardiography
* Indication of surgical aortic valve replacement for AS: will be defined in each center in accordance with ESC guidelines.
* Patient ≥ 70 years old and NYHA class ≥2 and LVEF <60% or global LV strain more than "-17%".
* Written consent prior to surgery.

Exclusion Criteria:

* Other severe disease with a life prognosis below than 1 year.
* Already known other causes of amyloidosis than senile amyloidosis will be excluded.
* Patients unsuitable for AS surgery as defined by ESC guidelines 2012.
* Significant mitral valve disease needing a surgical treatment.
* Significant aortic regurgitation (class >III).

NB: Patients with pacemaker will be included but will not perform the cardiac MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical composite criterion: All causes of death and cardiovascular hospitalization at 1 year after surgery | 1 year
  All causes of death and cardiovascular hospitalization at 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud DAMY, MD PhD, Principal Investigator — CHU Henri Mondor, Paris
Locations (5):
- France (5):
  - CHU d'Amiens, Amiens
  - Hôpital Henri Mondor, Créteil
  - Chu Rennes, Rennes
  - Centre Cardiologique du Nord, Saint-Denis
  - CHU de Toulouse, Toulouse